CLINICAL TRIAL: NCT04266860
Title: Establishing Clinical Utility of a New Diagnostic Test for Rheumatology Patients: A CPV® Randomized Controlled Trial
Brief Title: Establishing Clinical Utility of a New Diagnostic Test for Rheumatology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: DxTerity Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01DXT2019
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Lupus Nephritis; Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study will enroll practicing rheumatologists in the US, who will be randomly assigned to either an intervention or control arm.
  All eligible and consented participants will complete two rounds of three patient simulations.
  The intervention arm only will receive educational material about the DxTerity test in between these two rounds, and be provided simulated DxTerity test results in the second round of simulated cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental-arm providers will complete two rounds of three simulated patient cases (CPVs) with two additions described in the next column:
  Interventions: Other: Experimental - Test Results and Education
- Control (No Intervention): These providers will complete two rounds of three simulated patient cases (CPVs) only.

INTERVENTIONS:
Other: Experimental - Test Results and Education — First, these providers will receive educational materials (e.g. a slide deck, mock test result and one-page fact sheet) meant to mimic what physicians will receive in the real-world market as they learn about the DxTerity test.
  Second, within each of their second-round cases, intervention-arm physicians only will receive simulated test results from the DxTerity test at the clinically-appropriate point in each case.
  Arms: Experimental

SUMMARY:
This study will collect high-quality randomized controlled data from a nationally representative sample of practicing rheumatologists to determine how they currently manage patients with SLE (systemic lupus erythematosus) and how the results of DxTerity's IFN-1 (interferon type I) test change clinical decision making.

DETAILED DESCRIPTION:
This study will collect high-quality randomized controlled data from a nationally representative sample of practicing rheumatologists to determine how they currently manage patients with SLE and how the results of the IFN-1 test change clinical decision making. Data from this study will better illuminate the clinical use cases in which the IFN-1 test has the most significant impact on clinical decision making (and thus the largest clinical utility) and the associated physician characteristics (e.g., age, practice setting, training) associated with test adoption.

This study leverages simulated patient cases, called Clinical Performance and Value vignettes (CPVs), in a proven methodology to rapidly measure physician care decisions. CPVs are a unique and scalable tool that standardizes practice measurement by having all providers care for the same (virtual) patients. With all providers caring for the same patients, the CPVs generate unbiased data that yields powerful insights into clinical decision making and how these decisions change with the introduction of a new product or solution. CPVs have been validated and used effectively in rheumatology. Data from the CPVs can quickly demonstrate the clinical utility of a solution, be published in peer-reviewed literature, inform marketing strategies and positively impact coverage and reimbursement decisions.

The study is a prospective cohort trial with six steps:

1. Enrollment: The study will enroll an estimated 166 practicing rheumatologists who practice in the U.S. and are determined to be eligible by an eligibility screener.
2. Provider survey: Once providers are enrolled in the study, they will be asked to complete a questionnaire describing their practice and professional background.
3. Randomization: The 166 rheumatologists will be randomized into equally-sized control and intervention arms.
4. CPVs (First Round): Physicians will complete three randomly-assigned CPV patient simulations. Cases will be identical across the intervention and control arms. All interactive cases are presented on an online platform, and are accessible via unique weblinks and any internet-connected computer.
5. Intervention education: Intervention-arm rheumatologists will receive educational materials describing the clinical validation and use cases of the IFN-1 test. This material will replicate what physicians would receive as part of an actual marketing push introducing them to the IFN-1 test. These materials may be comprised of a slide deck, fact sheet, webinar, and/or case studies.
6. CPVs (Second Round): Physicians will then complete three additional CPV patient simulations in random order. Cases will be identical across the intervention and control arms, except that the intervention arm will receive IFN-1 test results at an appropriate point in each simulated case in the post-intervention round. Control arm physicians will continue to have access to standard of care diagnostic tools only.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified in rheumatology for at least two years
2. Averaging at least 20 hours per week of clinical and patient care duties over the last six months
3. Practicing in the U.S.
4. English speaking
5. Access to the internet
6. Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

1. Non-English speaking
2. Practicing in an academic setting
3. Unable to access the internet
4. Not practicing in the U.S.
5. Not averaging at least 20 hours per week of clinical or patient care duties over the last six months
6. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
CPV-measured pre-/post-score difference | 2-4 weeks
  Doctors receive scores on their simulated cases, or CPVs, based upon their quality of care. This measure will assess the pre- vs post-difference in the overall and the diagnostic and treatment quality scores between control physicians using standard of care diagnostic tools and intervention physicians with access to DxTerity test results, including by use case types.
CPV-measured value of care | 2-4 weeks
  Doctors make decisions in their simulated cases, or CPVs, including which tests and/or treatments to order for their virtual patients. This measure will model whether using IFN-1 results in higher-value care decisions in these CPV cases, including more appropriate use of disease modifying agents, for lupus-related care in different use cases.

SECONDARY OUTCOMES:
CPV-measured baseline variation | 1 week
  Doctors receive scores on their simulated cases, or CPVs, based upon their quality of care. This measure will assess the baseline levels of score variation in the work-up and management of lupus patients among all participants, including by use case types

CONTACTS AND LOCATIONS:
Overall Officials: John Peabody, MD, PhD, Principal Investigator — President, QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgon TB, Cox-Chapman J, Czarnecki C, Kropp R, Guerriere R, Paculdo D, Peabody JW. Engaging Primary Care Providers to Reduce Unwanted Clinical Variation and Support ACO Cost and Quality Goals: A Unique Provider-Payer Collaboration. Popul Health Manag. 2019 Aug;22(4):321-329. doi: 10.1089/pop.2018.0111. Epub 2018 Oct 17. PMID 30328782
- [Background] Peabody J, Martin M, DeMaria L, Florentino J, Paculdo D, Paul M, Vanzo R, Wassman ER, Burgon T. Clinical Utility of a Comprehensive, Whole Genome CMA Testing Platform in Pediatrics: A Prospective Randomized Controlled Trial of Simulated Patients in Physician Practices. PLoS One. 2016 Dec 30;11(12):e0169064. doi: 10.1371/journal.pone.0169064. eCollection 2016. PMID 28036350
- [Background] Peabody JW, Strand V, Shimkhada R, Lee R, Chernoff D. Impact of rheumatoid arthritis disease activity test on clinical practice. PLoS One. 2013 May 7;8(5):e63215. doi: 10.1371/journal.pone.0063215. Print 2013. PMID 23667587
- [Background] Solon O, Woo K, Quimbo SA, Shimkhada R, Florentino J, Peabody JW. A novel method for measuring health care system performance: experience from QIDS in the Philippines. Health Policy Plan. 2009 May;24(3):167-74. doi: 10.1093/heapol/czp003. Epub 2009 Feb 18. PMID 19224955
- [Background] DeMaria L, Acelajado MC, Luck J, Ta H, Chernoff D, Florentino J, Peabody JW. Variations and practice in the care of patients with rheumatoid arthritis: quality and cost of care. J Clin Rheumatol. 2014 Mar;20(2):79-86. doi: 10.1097/RHU.0000000000000076. PMID 24561410
- [Background] Peabody JW, Luck J, Glassman P, Jain S, Hansen J, Spell M, Lee M. Measuring the quality of physician practice by using clinical vignettes: a prospective validation study. Ann Intern Med. 2004 Nov 16;141(10):771-80. doi: 10.7326/0003-4819-141-10-200411160-00008. PMID 15545677